CLINICAL TRIAL: NCT06278454
Title: A Phase I Study to Evaluate the Safety, Tolerance and Efficacy of NRT6008 Injection in Unresectable Locally Advanced Pancreatic Cancer (LAPC)
Brief Title: Safety and Efficacy of NRT6008 in Patients With Unresectable Locally Advanced Pancreatic Cancer (LAPC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu New Radiomedicine Technology Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NrtPac-1; CTR20240312 (Other: Center for Drug Evaluation, NMPA)
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: Yttrium-90; Endoscopic ultrasound-guided fine-needle injection; Locally Advanced Pancreatic Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NRT6008 Injection (Experimental): In this study, participants shall receive NRT6008 injection in combination with chemotherapy.
  Interventions: Drug: NRT6008 Injection + Systematic chemotherapy

INTERVENTIONS:
Drug: NRT6008 Injection + Systematic chemotherapy — -Systematic chemotherapy The chemotherapy regimen is selected by the investigators at the consideration of participants' conditions, with either GN or (m)FOLFIRINOX.
  GN: gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2, every 21 days (3 weeks/cycle).
  FOLFIRINOX: oxaliplatin 85 mg/m^2, irinotecan 180 mg/m^2, leucovorin 400 mg/m^2 and fluorouracil 400 mg/m^2 given as a bolus followed by 2400 mg/m^2 given as a 46-hour continuous infusion, every 2 weeks (4 weeks/cycle).
  mFOLFIRINOX: oxaliplatin 85 mg/m^2, irinotecan 180 mg/m^2, leucovorin 400 mg/m^2, and fluorouracil 2400 mg/m^2 given as a 46-hour continuous infusion, every 2 weeks (4 weeks/cycle).
  -NRT6008 injection administration: NRT6008 injection is implanted into pancreatic tumor via endoscopic ultrasound (EUS)-guided fine-needle injection, at the instruction of the investigator. The dose of NRT6008 injection is determined by tumor volume and selected tumor average absorbed dose.
  Other Names: Investigational Product + Systematic chemotherapy

SUMMARY:
This is a single arm, open label, multi-center phase I study, including phase Ia dose escalation and phase Ib dose expansion. Safety review committee (SRC) will be formed to monitor safety and efficacy data through the study. And the independent review committee (IRC) will be formed to monitor efficacy data through the study.

DETAILED DESCRIPTION:
The efficacy and safety of Yttrium-90 carbon microspheres in patients with unresectable LAPC remain unknown. This trial is a prospective, multicenter, open-label, single-arm phase I trial designed to evaluate the safety and efficacy of NRT6008 injection. The primary objective is to evaluate the safety of NRT6008 Injection. While the secondary objectives include the assessments of the preliminary efficacy. In addition, the distribution of NRT6008 injection in human body, and the changes of tumor biomarkers and the improvement of cancer pain status of participants after administration will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤80 years, able to comprehend and sign an informed consent form;
2. Diagnosed with pancreatic adenocarcinoma confirmed histologically or cytologically;
3. Evaluated as unresectable LAPC by the investigator, or having contraindications to surgery, or refusing surgical resection (only patients with non-regional lymph node metastasis are eligible);
4. ECOG performance status score ≤1;
5. Expected survival ≥3 months;
6. According to RECIST v1.1 criteria, there is only one measurable lesion in the pancreas confirmed by imaging, and the lesion has the shortest axis diameter ≥2.0 cm, the longest axis diameter ≤6.0 cm (based on baseline imaging);
7. Adequate normal organ and marrow function as defined below: (1) Renal function: serum creatinine ≤1.5×ULN, or creatinine clearance ≥60 mL/min (calculated by the Cockcroft-Gault formula); (2) Liver function: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3×ULN; serum total bilirubin ≤1.5×ULN; (3) Bone marrow function [[no blood transfusion or granulocyte colony-stimulating factor (G-CSF), human thrombopoietin (TPO), or TPO receptor agonist treatment within 14 days prior to signing informed consent]: neutrophils ≥1.5×10^9/L, hemoglobin ≥90 g/L, platelets ≥100×10^9/L; (4) Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
8. Female and male participants of reproductive age must voluntarily agree to practice strict and effective contraception after signing the informed consent form, during the study period, and within 12 months after administration of the investigational drug. Males are prohibited from donating sperm during this period. Female participants of reproductive age must have a negative pregnancy test result during the screening period and within 24 hours before administration of the investigational drug.

Exclusion Criteria:

1. Allergic to the investigational drug NRT6008 injection itself or any of its components;
2. Contraindications to any of the three optional systemic chemotherapy regimens in this study judged by investigators;
3. Previous anti-tumor treatments for pancreatic cancer, including but not limited to chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc. Except for discontinuation of traditional chinese medicine or herbal medicine for at least 7 days prior to the screening period;
4. Contraindications to anesthesia;
5. History of any other malignant tumors within 5 years before receiving investigational drug treatment, except for cases of cured non-melanoma skin cancer, cervical carcinoma in situ, or basal cell carcinoma of the skin, Stage I Grade 1 endometrial carcinoma, or thyroid cancer;
6. Presence or suspected presence of distant metastases according to imaging;
7. Pregnant or lactating females;
8. Participants assessed by the investigators to be at high risk or had difficulty in operation for EUS-FNI procedures;
9. Evidence of radiographic invasion into stomach, duodenum or peritoneum;
10. Participants with chronic diseases that are actively treated but not well controlled, such as primary hypertension, diabetes, etc.;
11. Within 6 months prior to the the first administration of chemotherapy, occurrence of acute pancreatitis, severe gastrointestinal bleeding, severe cardiovascular diseases (including but not limited to stroke, unstable angina), or occurrence of acute infections requiring systemic treatment within 2 weeks before the screening period;
12. Participated in other interventional clinical trials within 1 month prior to the first administration of chemotherapy;
13. Positive for human immunodeficiency virus (HIV) antibodies;
14. Positive for hepatitis B virus (HBV) surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb), HBV DNA testing required, participants with HBV-DNA levels below the lower limit of the reference range or < 500 IU/mL will be eligible for inclusion in this study (use of antiviral drugs during the study period is required);
15. Positive for hepatitis C virus (HCV) antibodies, HCV RNA testing required, participants with negative HCV RNA results will be eligible for inclusion in this study;
16. Participants with syphilis infection or active tuberculosis;
17. Other reasons deemed unsuitable for participation in this trial by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or the recommended phase Ⅱ dose (RP2D) | 28 days after NRT6008 administration
  Optimal dose for NRT6008 injection
Dose-limiting toxicity (DLT) | 28 days after NRT6008 administration
  Incidence rate of DLT
Adverse events (AE) and severe adverse events (SAE) | Up to 52 weeks
  Incidence rate and severity of AE and SAE

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 52 weeks
  According to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, version 1.1 (evaluated by the investigator and Independent Review Committee respectively)
Duration of response (DOR) | Up to 52 weeks
  According to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, version 1.1 (evaluated by the investigator and Independent Review Committee respectively)
Progression-free survival (PFS) | Up to 52 weeks
  According to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, version 1.1 (evaluated by the investigator and Independent Review Committee respectively)
Overall survival (OS) | Up to 52 weeks
  How long the participant lives after the administration
Resection rate (R0 and R1) | Up to 52 weeks
  R0 (≥1 mm margin), R1 (<1 mm clearance)

OTHER OUTCOMES:
Concentration of tumor biomarkers | Up to 52 weeks
  Changes of tumor biomarkers through the study
Numeric rating scale (NRS) of pain | Up to 52 weeks
  Changes of Numeric rating scale (NRS) score. Patients should choose from 4 main categories, totaling 11 scores (0-10): namely no pain (0), mild pain (1-3), moderate pain (4-6), severe pain (7-10). As the score increases, the intensity of pain also rises.
Distribution of NRT6008 injection in human body and radioactivity of biological samples | Up to 48 hours
  Distribution of NRT6008 injection in human body and radioactivity of Yttrium-90 in blood, urine, and feces (if available)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Principal Investigator — Changhai Hospital
Locations (6):
- China (6):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Chongqing University Cancer Hospital, Chongqing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No